CLINICAL TRIAL: NCT00393692
Title: Prospective Natural History Study of Fundus Autofluorescence Imaging in Age-related Macular Degeneration (FAM-Study) Using Confocal Scanning Laser Ophthalmoscopy
Brief Title: Fundus Autofluorescence Imaging in Age-related Macular Degeneration Using Confocal Scanning Laser Ophthalmoscopy
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Frank G. Holz, Prof. Dr. med., University Hospital, Bonn
Other Study IDs: FAM-Study; DFG Priority Program AMD; SPP 1088; Ho 1926/1-3; Ho 1926/3-1; Ma 1723/1-1
Record Dates: First submitted 2006-10-26; First posted 2006-10-30 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Age-related Macular Degeneration
Keywords: Age-related macular degeneration; Geographic atrophy; drusen
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to define phenotypic variations in atrophic Age-Related Macular Degeneration (AMD) and to identify predictive factors for disease progression based on fundus autofluorescence imaging.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is the leading cause of legal blindness in the industrialized world beyond 50 years of age. Ageing changes of the retinal pigment epithelium (RPE) play a key role in the pathogenesis of the disease. In postmitotic RPE cells autofluorescent lipofuscin granules accumulate with age in the lysosomal compartment mainly as a byproduct of constant phagocytosis of membranous disks shed from photoreceptor outer segments. With the advent of confocal scanning laser ophthalmoscopy fundus autofluorescence mediated by RPE-lipofuscin accumulation can be visualized in vivo: We plan to identify fundus autofluorescence changes as predictive factors for the development of late stage manifestations and their variation over time. Furthermore, we plan to determine the effect of increased focal accumulations of autofluorescent material on retinal sensitivity using fundus perimetry. Examination of human donor eyes with AMD will allow for correlation of fundus autofluorescence alterations in vivo and in vitro. These investigations will be performed not only to better understand the role of lipofuscin accumulation in AMD but also to manipulate these mechanisms for both experimental and therapeutic ends.

ELIGIBILITY:
Inclusion Criteria:

* Must be considered reliable, willing and able to give informed consent.
* Age >50 years (male or female)
* Must have age-related macular degeneration in at least one eye
* Clear media to allow imaging

Exclusion Criteria:

* any history of retinal surgery, including laser treatment, photodynamic therapy, radiation or intravitreal injections
* history of retinal vascular occlusions
* any concurrent intraocular condition that, in the opinion of the investigator, could exclude the patient from the medical or ethical point of view

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with unilateral or bilateral geographic atrophy due to AMD, aged 50 years and older. German population
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2000-08; Primary Completion 2016-04 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Change of geographic atrophy size to baseline | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Frank G Holz, MD, Principal Investigator — University of Bonn
Locations (7):
- Germany (7):
  - Department of Ophthalmology, University of Aachen, Aachen
  - Department of Ophthalmology, University of Heidelberg, Heidelberg
  - Institute for Medical Statistics and Biometry, University of Heidelberg, Heidelberg
  - Department of Ophthalmology, University of Leipzig, Leipzig
  - • Institute for Biometry and Epidemiology, Ludwig-Maximilians-University, Munich
  - St. Franziskus Hospital Münster, Münster
  - Department of Ophthalmology, University of Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Holz FG, Bellmann C, Margaritidis M, Schutt F, Otto TP, Volcker HE. Patterns of increased in vivo fundus autofluorescence in the junctional zone of geographic atrophy of the retinal pigment epithelium associated with age-related macular degeneration. Graefes Arch Clin Exp Ophthalmol. 1999 Feb;237(2):145-52. doi: 10.1007/s004170050209. PMID 9987631
- [Background] Holz FG, Bellman C, Staudt S, Schutt F, Volcker HE. Fundus autofluorescence and development of geographic atrophy in age-related macular degeneration. Invest Ophthalmol Vis Sci. 2001 Apr;42(5):1051-6. PMID 11274085
- [Background] Schmitz-Valckenberg S, Fleckenstein M, Scholl HP, Holz FG. Fundus autofluorescence and progression of age-related macular degeneration. Surv Ophthalmol. 2009 Jan-Feb;54(1):96-117. doi: 10.1016/j.survophthal.2008.10.004. PMID 19171212
- [Background] Fleckenstein M, Charbel Issa P, Helb HM, Schmitz-Valckenberg S, Scholl HP, Holz FG. Correlation of lines of increased autofluorescence in macular dystrophy and pigmented paravenous retinochoroidal atrophy by optical coherence tomography. Arch Ophthalmol. 2008 Oct;126(10):1461-3. doi: 10.1001/archopht.126.10.1461. No abstract available. PMID 18852430
- [Background] Schmitz-Valckenberg S, Fleckenstein M, Gobel AP, Sehmi K, Fitzke FW, Holz FG, Tufail A. Evaluation of autofluorescence imaging with the scanning laser ophthalmoscope and the fundus camera in age-related geographic atrophy. Am J Ophthalmol. 2008 Aug;146(2):183-92. doi: 10.1016/j.ajo.2008.04.006. Epub 2008 Jun 2. PMID 18514607
- [Result] Schmitz-Valckenberg S, Bindewald-Wittich A, Dolar-Szczasny J, Dreyhaupt J, Wolf S, Scholl HP, Holz FG; Fundus Autofluorescence in Age-Related Macular Degeneration Study Group. Correlation between the area of increased autofluorescence surrounding geographic atrophy and disease progression in patients with AMD. Invest Ophthalmol Vis Sci. 2006 Jun;47(6):2648-54. doi: 10.1167/iovs.05-0892. PMID 16723482
- [Result] Bindewald A, Schmitz-Valckenberg S, Jorzik JJ, Dolar-Szczasny J, Sieber H, Keilhauer C, Weinberger AW, Dithmar S, Pauleikhoff D, Mansmann U, Wolf S, Holz FG. Classification of abnormal fundus autofluorescence patterns in the junctional zone of geographic atrophy in patients with age related macular degeneration. Br J Ophthalmol. 2005 Jul;89(7):874-8. doi: 10.1136/bjo.2004.057794. PMID 15965170
- [Result] Deckert A, Schmitz-Valckenberg S, Jorzik J, Bindewald A, Holz FG, Mansmann U. Automated analysis of digital fundus autofluorescence images of geographic atrophy in advanced age-related macular degeneration using confocal scanning laser ophthalmoscopy (cSLO). BMC Ophthalmol. 2005 Apr 6;5:8. doi: 10.1186/1471-2415-5-8. PMID 15813972
- [Result] Schmitz-Valckenberg S, Bultmann S, Dreyhaupt J, Bindewald A, Holz FG, Rohrschneider K. Fundus autofluorescence and fundus perimetry in the junctional zone of geographic atrophy in patients with age-related macular degeneration. Invest Ophthalmol Vis Sci. 2004 Dec;45(12):4470-6. doi: 10.1167/iovs.03-1311. PMID 15557456
- [Result] Schmitz-Valckenberg S, Jorzik J, Unnebrink K, Holz FG; FAM Study Group. Analysis of digital scanning laser ophthalmoscopy fundus autofluorescence images of geographic atrophy in advanced age-related macular degeneration. Graefes Arch Clin Exp Ophthalmol. 2002 Feb;240(2):73-8. doi: 10.1007/s00417-001-0413-3. PMID 11933894
- [Result] Dreyhaupt J, Mansmann U, Pritsch M, Dolar-Szczasny J, Bindewald A, Holz FG. Modelling the natural history of geographic atrophy in patients with age-related macular degeneration. Ophthalmic Epidemiol. 2005 Dec;12(6):353-62. doi: 10.1080/09286580591005723. PMID 16283987
- [Result] Bindewald A, Bird AC, Dandekar SS, Dolar-Szczasny J, Dreyhaupt J, Fitzke FW, Einbock W, Holz FG, Jorzik JJ, Keilhauer C, Lois N, Mlynski J, Pauleikhoff D, Staurenghi G, Wolf S. Classification of fundus autofluorescence patterns in early age-related macular disease. Invest Ophthalmol Vis Sci. 2005 Sep;46(9):3309-14. doi: 10.1167/iovs.04-0430. PMID 16123434
- [Result] Einbock W, Moessner A, Schnurrbusch UE, Holz FG, Wolf S; FAM Study Group. Changes in fundus autofluorescence in patients with age-related maculopathy. Correlation to visual function: a prospective study. Graefes Arch Clin Exp Ophthalmol. 2005 Apr;243(4):300-5. doi: 10.1007/s00417-004-1027-3. Epub 2004 Oct 13. PMID 15864618
- [Result] Bellmann C, Jorzik J, Spital G, Unnebrink K, Pauleikhoff D, Holz FG. Symmetry of bilateral lesions in geographic atrophy in patients with age-related macular degeneration. Arch Ophthalmol. 2002 May;120(5):579-84. doi: 10.1001/archopht.120.5.579. PMID 12003606
- [Derived] Pfau M, Lindner M, Goerdt L, Thiele S, Nadal J, Schmid M, Schmitz-Valckenberg S, Sadda SR, Holz FG, Fleckenstein M; Fundus Autofluorescence in Age-Related Macular Degeneration Study Group. PROGNOSTIC VALUE OF SHAPE-DESCRIPTIVE FACTORS FOR THE PROGRESSION OF GEOGRAPHIC ATROPHY SECONDARY TO AGE-RELATED MACULAR DEGENERATION. Retina. 2019 Aug;39(8):1527-1540. doi: 10.1097/IAE.0000000000002206. PMID 29781974
- [Derived] Lindner M, Kosanetzky S, Pfau M, Nadal J, Gordt LA, Schmitz-Valckenberg S, Schmid M, Holz FG, Fleckenstein M; FAM-Study Group. Local Progression Kinetics of Geographic Atrophy in Age-Related Macular Degeneration Are Associated With Atrophy Border Morphology. Invest Ophthalmol Vis Sci. 2018 Mar 20;59(4):AMD12-AMD18. doi: 10.1167/iovs.17-23203. PMID 29558533
- [Derived] Lindner M, Nadal J, Mauschitz MM, Luning A, Czauderna J, Pfau M, Schmitz-Valckenberg S, Holz FG, Schmid M, Fleckenstein M. Combined Fundus Autofluorescence and Near Infrared Reflectance as Prognostic Biomarkers for Visual Acuity in Foveal-Sparing Geographic Atrophy. Invest Ophthalmol Vis Sci. 2017 May 1;58(6):BIO61-BIO67. doi: 10.1167/iovs.16-21210. PMID 28475704
- [Derived] Lindner M, Boker A, Mauschitz MM, Gobel AP, Fimmers R, Brinkmann CK, Schmitz-Valckenberg S, Schmid M, Holz FG, Fleckenstein M; Fundus Autofluorescence in Age-Related Macular Degeneration Study Group. Directional Kinetics of Geographic Atrophy Progression in Age-Related Macular Degeneration with Foveal Sparing. Ophthalmology. 2015 Jul;122(7):1356-65. doi: 10.1016/j.ophtha.2015.03.027. Epub 2015 May 9. PMID 25972258
- [Derived] Fleckenstein M, Schmitz-Valckenberg S, Lindner M, Bezatis A, Becker E, Fimmers R, Holz FG; Fundus Autofluorescence in Age-Related Macular Degeneration Study Group. The "diffuse-trickling" fundus autofluorescence phenotype in geographic atrophy. Invest Ophthalmol Vis Sci. 2014 May 2;55(5):2911-20. doi: 10.1167/iovs.13-13409. PMID 24699379
- [Derived] Smailhodzic D, Fleckenstein M, Theelen T, Boon CJ, van Huet RA, van de Ven JP, Den Hollander AI, Schmitz-Valckenberg S, Hoyng CB, Weber BH, Holz FG, Klevering BJ. Central areolar choroidal dystrophy (CACD) and age-related macular degeneration (AMD): differentiating characteristics in multimodal imaging. Invest Ophthalmol Vis Sci. 2011 Nov 21;52(12):8908-18. doi: 10.1167/iovs.11-7926. PMID 22003107
- [Derived] Fleckenstein M, Schmitz-Valckenberg S, Adrion C, Visvalingam S, Gobel AP, Mossner A, von Strachwitz CN, Mackensen F, Pauleikhoff D, Wolf S, Mansmann U, Holz FG; FAM Study Group. Progression of age-related geographic atrophy: role of the fellow eye. Invest Ophthalmol Vis Sci. 2011 Aug 22;52(9):6552-7. doi: 10.1167/iovs.11-7298. PMID 21757586
- [Derived] Fleckenstein M, Schmitz-Valckenberg S, Martens C, Kosanetzky S, Brinkmann CK, Hageman GS, Holz FG. Fundus autofluorescence and spectral-domain optical coherence tomography characteristics in a rapidly progressing form of geographic atrophy. Invest Ophthalmol Vis Sci. 2011 Jun 1;52(6):3761-6. doi: 10.1167/iovs.10-7021. PMID 21310912
- [Derived] Schmitz-Valckenberg S, Fleckenstein M, Gobel AP, Hohman TC, Holz FG. Optical coherence tomography and autofluorescence findings in areas with geographic atrophy due to age-related macular degeneration. Invest Ophthalmol Vis Sci. 2011 Jan 5;52(1):1-6. doi: 10.1167/iovs.10-5619. PMID 20688734
- [Derived] Fleckenstein M, Schmitz-Valckenberg S, Adrion C, Kramer I, Eter N, Helb HM, Brinkmann CK, Charbel Issa P, Mansmann U, Holz FG. Tracking progression with spectral-domain optical coherence tomography in geographic atrophy caused by age-related macular degeneration. Invest Ophthalmol Vis Sci. 2010 Aug;51(8):3846-52. doi: 10.1167/iovs.09-4533. Epub 2010 Mar 31. PMID 20357194
- [Derived] Fleckenstein M, Adrion C, Schmitz-Valckenberg S, Gobel AP, Bindewald-Wittich A, Scholl HP, Mansmann U, Holz FG; FAM Study Group. Concordance of disease progression in bilateral geographic atrophy due to AMD. Invest Ophthalmol Vis Sci. 2010 Feb;51(2):637-42. doi: 10.1167/iovs.09-3547. Epub 2009 Sep 24. PMID 19797219
- See also: German Research Council — http://www.dfg.de/en